CLINICAL TRIAL: NCT05781438
Title: Feasibility of an In-home Standing and Walking Intervention for Infants With and at High Risk of Cerebral Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: California Physical Therapy Association (Unknown); Cerebral Palsy Foundation (Unknown)
Responsible Party: Principal Investigator, Barbara Sargent, Associate Professor of Clinical Physical Therapy, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UP-22-00866
Record Dates: First submitted 2022-12-31; First posted 2023-03-23 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Cerebral Palsy
Keywords: Infant
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Single-subject research design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- In-home standing and walking intervention (Experimental): Infants will participate in the in-home standing and walking intervention for 16 weeks. In addition, infants will continue with any intervention in the community recommended by their health care team.
  Interventions: Behavioral: In-home standing and walking intervention

INTERVENTIONS:
Behavioral: In-home standing and walking intervention — Parents/legal guardians will be educated on and provided an activity booklet on intensive standing and walking play activities for their infant in a 9 by 9 foot body-weight support system (BWS). Activities include: squatting play at a couch or table, cruising along and between furniture, walking with a push toy or with one or two hands held, walking without support, and kicking and throwing a soft ball.
  For 16 weeks, parents/legal guardians will be encouraged to implement the parent-led, intensive standing and walking intervention using BWS for at least 5 days/week for 30-60 min/day, with weekly telehealth calls and monthly home visits to coach parents in identifying key activities and progressing the program.

SUMMARY:
The purpose of this study is to evaluate the feasibility and begin to evaluate the effect of an intensive in-home standing and walking intervention for infants with or at high risk of cerebral palsy.

DETAILED DESCRIPTION:
Seventy percent of children with cerebral palsy (CP) will walk, yet walking occurs much later than typically-developing children and may require use of a walker or crutches. The walking impairment is caused by an early lesion to the motor areas of the brain which disrupts the formation of appropriate neural connections, specifically projections of the corticospinal tract from the motor cortex to spinal cord motor circuits. The critical period of lower extremity neuromotor development, when intervention is expected to be most effective, begins before 12 months of age with the establishment of appropriate spinal connections and extends to 2 years of age with the presence of mature myelin in the corticospinal tract at the lumbar level. Based on this research, we propose that to optimize future walking outcomes of individuals with CP, it is critical to promote standing and walking practice during infancy before the age of 12 months.

The purpose of this study is to evaluate the feasibility and begin to evaluate the effect of an intensive in-home standing and walking intervention for infants with or at high risk of CP. Eight infants with or at high risk of CP will enter the study at 5 to 12-months of age. All infants will participate in 3 conditions: 8-weeks no intervention baseline, 16-weeks intervention, and 8-weeks no intervention follow-up. During the intervention weeks, parents will implement the in-home intensive standing and walking intervention with body-weight support 5 days/week for 30-60 min/day, with weekly telehealth calls and monthly home visits to progress the program. The body-weight support system allows infants to independently explore a 9 by 9-foot space in standing without physical assist from their parents or other adults.

Outcomes will be measured at baseline, monthly throughout the 8 month study, and at 2 years of age. Feasibility of implementing the interventions will be assessed. Secondary outcomes will include standardized assessments of motor, cognitive, and language development of the infants.

ELIGIBILITY:
Inclusion Criteria:

* Infants with or at high risk of cerebral palsy (CP) who either:

  * have been diagnosed with CP by a medical professional, or
  * are at high risk of CP defined as having both:

    * clinical brain imaging indicating CP, such as (i) white matter injury (cystic periventricular leukomalacia or periventricular hemorrhagic infarctions), (ii) hypoxic-ischemic encephalopathy, or (iii) neonatal stroke, and
    * a score less than 63 or more than 5 asymmetries on the Hammersmith Infant Neurological Examination (HINE).

Exclusion Criteria:

* prenatal substance abuse,
* congenital malformations,
* drug-resistant epilepsy,
* visual impairment that hinders the infant from seeing toys,
* hearing impairment that hinders the infant from responding to sound,
* living in a location inaccessible by study personnel for in-home data collections,
* participant over 50 lbs in weight.

Ages: 5 Months to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Estimated)
Dates: Start 2023-03-26 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the in-home standing and walking intervention | 4 months
  Feasibility will be quantified by: parent survey of the: (a) infants' level of enjoyment during the intervention, (b) ease of use of the body-weight support system, (c) time participating in intervention, (d) time to put child in and take child out of the body-weight support, (e) perception of the effect of the intervention on the infant's motor skills, (f) perception of the effects of the intervention on the infant's non-motor skills (cognition, social, language), (g) overall perception of intervention as beneficial. The parent survey is on a likert scale from 1 to 5; a higher score denotes a better outcome.

SECONDARY OUTCOMES:
Bayley Scales of Infant and Toddler Development, 4th edition (Bayley-4) | 2 years
  The Bayley Scales of Infant and Toddler Development, 4th edition (Bayley-4) is a standardized developmental assessment that provides raw scores for 5 subtests (cognitive, expressive communication, receptive communication, fine motor, gross motor) and standard score norms converted to percentiles for 3 scales (cognition, communication, motor). The Bayley-4 raw scores range from 0-162 for the cognitive subtest, 0-84 for the receptive communication subtest, 0-74 for the expressive communication subtest, 0-92 for the fine motor subtest, and 0-116 for the gross motor subtest; a higher score denotes a better outcome. The Bayley-4 standard score norms are converted to percentiles from <0.1 to >99.9 for the cognitive, language, and motor scales; a higher percentile denotes a better outcome.
Gross Motor Function Measure (GMFM-88) | 2 years
  The Gross Motor Function Measure (GMFM-88) is a standardized motor assessment designed to assess gross motor function of children with cerebral palsy. The GMFM-88 raw scores range from 0-51 for the lying and rolling subtest, 0-60 for the sitting subtest, 0-42 for the crawling and kneeling subtest, 0-39 for the standing subtest, and 0-72 for the walking, running and jumping subtest; a higher score denotes a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Sargent, PhD, PT, Principal Investigator — University of Southern California, Division of Biokinesiology and Physical Therapy
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No